CLINICAL TRIAL: NCT07094126
Title: Blood Pressure Monitor (KD-595) Clinical Test (Cuff Range: 15-24cm, 22-42cm, 40-48cm)
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Andon Health 14
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject use both KD-595 Blood Pressure Monitor and mercury sphygmomanometers

SUMMARY:
The purpose of this study is to verify the accuracy of the three (3) cuffs with blood pressure monitor device.

ELIGIBILITY:
Inclusion Criteria:

* Normal blood pressure and hypertensive patients over 12 years old

Exclusion Criteria:

* Patients with serious arrhythmias or a high frequency of arrhythmias
* Pregnant woman
* Other investigators believe that it is not suitable to participate in this clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Normal blood pressure and hypertensive patients over 12 years old
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2023-10-08 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Monitor Accuracy | 30 minutes
  All the test results of the electronic blood pressure monitor with three (3) cuffs is within the accuracy creteria, with the merury sphygmomanometer as control

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, the Air Force Medical University, Xi’an, Shanxi, China